CLINICAL TRIAL: NCT06514898
Title: MATCHPOINT - Medulloblastoma Adoptive T Cell Therapy, DC Vaccines, and Hematopoietic Stem Cells Combined With Immune checkPOINT Blockade
Brief Title: Adoptive T Cell Therapy, DC Vaccines, and Hematopoietic Stem Cells Combined With Immune checkPOINT Blockade in Patients With Medulloblastoma
Acronym: MATCHPOINT
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202400861-A; OCR45772 (Other: University of Florida)
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Group 3 Medulloblastoma; Recurrent Group 4 (Non-SHH/Non-WNT) Medulloblastoma
MeSH Terms: conditions — Medulloblastoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Diphtheria-Tetanus Vaccine; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adoptive Cellular Therapy (ACT) + PD-1 blockade with pembrolizumab (Experimental): ACT + PD-1 blockade consists of the intravenous delivery of ex vivo expanded tumor-reactive lymphocytes and autologous hematopoietic stem cells (HSCs) with concomitant tumor RNA-pulsed DC vaccines followed by intravenous delivery of PD-1 blocking antibodies.
  Interventions: Biological: TTRNA-DC vaccines with GM-CSF; Biological: TTRNA-xALT; Drug: Td vaccine; Biological: autologous HSCs; Drug: Pembrolizumab

INTERVENTIONS:
Biological: TTRNA-DC vaccines with GM-CSF — After chemoradiation subjects will receive the first cycle of dose-intensified TMZ followed by three biweekly TTRNA-DC vaccines with GM-CSF. Monthly DC vaccines will be given during TMZ Cycles 2-5 for Groups A and B and 48-96 hours after completion of TMZ Cycle 6 Day 21 for Group A and 12-36 hours after HSCs for Group B. All subjects will receive an additional two bi-weekly vaccines during Cycle 6 for a total of 10 DC vaccines. All DC vaccines will be embedded with GM-CSF (150 µg per injection) and given intradermal.
  up to 9 intradermal DC vaccines (three -bi-weekly (q2 weeks) for priming, monthly for additional 2-3 cycles during T cell expansion, and three bi-weekly during T cell engraftment)
Biological: TTRNA-xALT — All participants will receive a single infusion of T-cells.
Drug: Td vaccine — A full Td booster vaccine will be administered IM at Vaccine #1 to all subjects, and vaccine site pretreatment will be administered to all subjects prior to Vaccine#3, #5, #7 and #9.
Biological: autologous HSCs — All participants will receive a single intravenous infusion of autologous HSCs.
Drug: Pembrolizumab — Participants will receive PD-1 blockade IV starting with ACT continuing for up to 2 years as long as tolerable and without disease progression.

SUMMARY:
This is a pilot study in a small number of children and young adults with relapsed/progressive medulloblastoma (MB) looking at the feasibility and safety of adoptive cell therapy plus PD-1 blockade.

DETAILED DESCRIPTION:
This is a single-site, single arm, unblinded, uncontrolled pilot study to evaluate the feasibility and safety of ACT + PD-1 blockade in children and young adults with suspected recurrence/progression of Group 3 or 4 (non-SHH/non-WNT) medulloblastoma since completion of definitive focal +/- craniospinal irradiation who are a candidate for surgical resection or biopsy.

After a screening consent is obtained for the collection of tumor sample, subjects will undergo standard of care resection for tumor debulking or biopsy for confirmatory diagnosis of disease progression. Tumor tissue will be collected during surgery for tumor debulking or biopsy for total tumor RNA and generation of investigational DC vaccine in parallel. Following biopsy and confirmatory pathologic diagnosis of recurrent MB, patients will be enrolled in the treatment phase of the trial after obtaining informed consent.

After surgery, patients will undergo a mobilized pheresis to collect PBMCs for DC generation and CD34+ HSCs. Amplified tumor RNA obtained from surgically resected or biopsied specimens will be used to generate total tumor RNA-pulsed DCs (TTRNA-DCs) manufactured while patients initiate post-surgical salvage chemotherapy regimen.

Salvage chemotherapy prescribed by treating neuro-oncologist will initiate 1-2 weeks after G-CSF mobilized leukapheresis for 1-3 cycles after which, treatment cycles will be paused, and the patients will receive 3 priming TTRNA-DCs vaccines every 2 weeks and undergo a non-mobilized leukapheresis to collect vaccine-boosted lymphocytes for ex vivo T cell expansion and generation of additional TTRNA-DC vaccines. Treatment with salvage chemotherapy will resume with monthly TTRNA-DC vaccines for an additional 1-3 cycles until ex vivo expanded T cells are manufactured and released from the UF cGMP facility.

For ACT, patients will undergo non-myeloablative conditioning with cyclophosphamide/fludarabine followed by infusion of ex vivo expanded tumor-reactive lymphocytes at 3 x 108 cells/Kg, infusion of autologous CD34+ HSCs (targeted dose of 2 x 106 CD34+ HSCs/Kg), PD-1 blockade and three biweekly intradermal TTRNA-DC vaccines to boost T cell engraftment and expansion.

The total immunotherapy regimen will consist of up to 9 intradermal DC vaccines (three -bi-weekly (q2 weeks) for priming, monthly for additional 2-3 cycles during T cell expansion, and three bi-weekly during T cell engraftment), a single intravenous infusion of ex vivo expanded tumor-reactive T cells, and a. single intravenous infusion of autologous HSCs; and PD-1 blockade IV starting with ACT continuing for up to 2 years as long as tolerable and without disease progression.

All patients will receive a full Td booster (5 Lf) IM vaccine 4-24 hours prior to Vaccine #1, regardless of booster history. All patients will undergo vaccine site pretreatment with a one-fifth dose of Td (1 Lf) intradermally, at the site of planned DC vaccine, 4-24 hours prior to vaccines #3, #5, #7 and #9.

ELIGIBILITY:
Inclusion Criteria:

1. Children and young adults age 4-30 years with suspected recurrence/progression of Group 3 or 4 (non-SHH/non-WNT) MB since completion of definitive focal +/- craniospinal irradiation who are a candidate for surgical resection or biopsy. Of the 6 evaluable subjects, a minimum of 3 slots must be reserved for patients with confirmed Group 4 MB. Patients who are unable to receive radiation therapy due to genetic disorders that put them at significant risk for radiation-induced secondary malignancies (i.e. Gorlin's syndrome or NF1 mutation) are eligible for enrollment at first disease recurrence/progression.
2. Must be a candidate for surgery/biopsy Or tumor tissue obtained clinically, has been previously stored in a biorepository suitable for tumor RNA extraction and amplification and sample is made available to the PI.
3. Karnofsky or Lansky Performance Status (KPS) ≥ 60% (KPS for > 16 years of age) or Lansky performance Score (LPS) of ≥ 60 (LPS for < 16 years of age)
4. Adequate bone marrow and organ function as defined below:

   * ANC ≥ 1,000/mcL (unsupported)
   * Platelets ≥ 100,000/mcL (unsupported for at least 3 days)
   * Hemoglobin ≥ 9 g/dL (may be supported)
   * Serum creatinine ≤ 1.5 x IULN OR Creatinine clearance by Cockcroft-Gault ≥ 60 mL/min for patients with serum creatinine > 1.5 x IULN
   * Serum total bilirubin ≤ 1.5 x IULN for age OR Direct bilirubin ≤ IULN for patients with total bilirubin > 1.5 x IULN for age
   * AST (SGOT) and ALT (SGPT) ≤ 3 x IULN for age
   * Cardiac shortening fraction ≥27% or LVEF ≥50% by echocardiogram
   * Adequate pulmonary function defined as baseline pulse oximetry of ≥92% on room air
5. For females of childbearing potential, negative serum pregnancy test at enrollment
6. For women of childbearing potential (WOCBP) must be willing to use acceptable contraceptive methods to avoid pregnancy throughout the study and for at least 24 weeks after the last dose of study drug.

   or For males with female partners of childbearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 24 weeks following the last dose of study drug.
7. Signed informed consent by patient and/or legally authorized representative

Exclusion Criteria:

this study:

1. Prior discontinuation of PD-1 inhibitor treatment due to toxicity or disease progression.
2. Corticosteroids equivalent to ≥ 4mg dexamethasone daily.
3. HIV, Hepatitis B, or Hepatitis C seropositive.
4. Known active infection or immunosuppressive disease.
5. Autoimmune disease requiring medical management with immunosuppressant.
6. Pregnancy or lactation, due to possible adverse effects on the developing fetus or infant.
7. Treatment with another investigational drug or other intervention within 30 days prior to projected first dose of study treatment (Priming phase with TTRNA-DC).
8. Severe, active co-morbidity, defined as follows:

   * Unstable angina and/or congestive heart failure requiring hospitalization.
   * Transmural myocardial infarction within the last 6 months.
   * Acute bacterial or fungal infection requiring intravenous antibiotics at time of enrollment.
   * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy.
   * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects.
   * Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
   * Major medical illnesses or psychiatric impairments that, in the investigator's opinion, will prevent administration or completion of protocol therapy.

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with immunotherapy-related dose-limiting toxicities after treatment with TTRNA-DCs, TTRNA-xALT and HSCs plus PD1 blockade | enrollment to completion of DLT window; up to 12 months
  Number of subjects with immunotherapy-related dose-limiting toxicities including 1) Grade III or greater non-neurologic toxicity; 2) Grade III neurologic toxicity that does not improve to Grade II or better within 5 days; or 3) Grade IV neurologic toxicity.
  For the purposes of evaluating the safety of ACT combined with PD-1 blockade, dose limiting toxicities will be assessed during the period beginning with administration of ex vivo expanded tumor-reactive (TTRNA- xALT) through 2 weeks post TTRNA -DC vaccine #9.
  Safety will be defined as < 1 DLT out of six enrolled and treated subjects.
Number of enrolled participants who receive qualified immunotherapy products out of the total number of participants enrolled. | enrollment up to 12 months
  Feasibility will be defined as capacity to enroll, manufacture, and administer qualified immunotherapy products (TTRNA-DCs, TTRNA-xALT and HSCs) to at least 66.7% of enrolled subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Duane Mitchell, MD, PhD, Study Chair — University of Florida; John Ligon, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Health, Gainesville, Florida, United States